CLINICAL TRIAL: NCT05371847
Title: Identifying Prognostic Variables for Persistent Upper Limb Dysfunctions After Breast Cancer Treatment: Longitudinal Cohort Study
Brief Title: Identifying Prognostic Variables for Persistent UL Dysfunctions After Breast Cancer Treatment -Reliability and Validity
Acronym: UPLIFT-BC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: KU Leuven (Other)
Collaborators: Universitaire Ziekenhuizen KU Leuven (Other); Vrije Universiteit Brussel (Other)
Responsible Party: Principal Investigator, An De Groef, Prof. Dr, KU Leuven
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: s66248-aim2
Record Dates: First submitted 2022-03-17; First posted 2022-05-12 (Actual); Last update posted 2024-05-01 (Actual); Status verified 2024-04

CONDITIONS: Breast Cancer
Keywords: upper limb dysfunction
MeSH Terms: conditions — Breast Neoplasms | interventions — Restraint, Physical

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- breast cancer patients (Active Comparator): Women and men in the prospective cohort study will be invited to participate in this additional validity and/or reliability testing
  Interventions: Other: assessment for upper limb dysfunction; Other: retest assessment
- healthy volunteers (Active Comparator): age- and gender-matched
  Interventions: Other: assessment for upper limb dysfunction; Other: retest assessment

INTERVENTIONS:
Other: assessment for upper limb dysfunction — clinical assessments and questionnaires
Other: retest assessment — For the test-retest reliability testing, participants will be invited to have an additional appointment approximately 1 week after the main assessment.

SUMMARY:
Breast cancer is the most frequently occurring cancer, assuming that it accounts for 29% of all new cancers in women (European Cancer Information System). The number of long-term survivors is increasing rapidly due to improving accuracy of the detecting methods, the early diagnosis and advances in cancer treatment.

The International Consortium for Health Outcomes Measurement Initiative described upper limb (UL) function as the health outcome that matters most for breast cancer survivors (BCS). 50% of BCS at 6 months post-radiotherapy suffer from of decreased UL function, i.e. difficulties in performing activities of daily living with the upper limb. Patients experiencing UL dysfunctions and other problems are less likely to be physically active. Given that physical inactivity is associated with an increased risk of mortality after breast cancer, taking away the barriers to physical activity (e.g. UL dysfunctions) is very important. Identifying these factors contributing to chronic UL dysfunction is important in terms of identifying targets for prospective evaluation and specific treatment approaches at specific time points during breast cancer treatment.

This study aims to find reliable and valid assessment methods for the prognostic factors and upper limb function itself in a small group of BCS and healthy volunteers.

ELIGIBILITY:
Inclusion Criteria for breast cancer patients

* Patients scheduled for surgery (mastectomy or breast conserving surgery; in combination with axillary lymph node dissection or sentinel node biopsy) for unilateral primary breast cancer or patients with oligometastatic breast cancer.
* Patients who receive adjuvant radiotherapy .
* Patients with a cognitive and language functioning enabling coherent Dutch communication between the examiner and the participant
* Patients who can comply with the protocol at baseline assessment and willing to provide written informed consent

Inclusion criteria healthy volunteers

* Healthy women and men(quickDASH<15) age- and gender-matched with a breast cancer patient from the main study
* Volunteers who can comply with the protocol at baseline assessment and willing to provide written informed consent

Exclusion Criteria breast cancer patients

* BCS with widespread distance metastases, previous breast surgery, or planned bilateral surgery
* And/or with a diagnosis of a neurological or rheumatological condition, diabetes,
* And/or BCS who are not available the entire duration of the study

Exclusion Criteria healthy volunteers

* History of breast cancer
* Patients with a diagnosis of neurological or rheumatological condition, diabetes

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2022-04-26 (Actual); Primary Completion 2025-02 (Estimated); Study Completion 2025-02 (Estimated)

PRIMARY OUTCOMES:
Reliability of measurements with MyotonPro | 1 week
  Inter- and intra-rater reliability will be tested. The MyotonPRO assessment for soft-tissue stiffness and elasticity will take place at the pectoralis major, upper trapezius, infraspinatus and teres major region, from which a mean stiffness index (N/m) will be calculated.
  approximately 1 week between test & retest
Validity of the evaluation tool for Myofascial Adhesions in Patients after Breast Cancer | 1 week
  The validity of the evaluation tool for Myofascial Adhesions in Patients after Breast Cancer (MAP-BC evaluation tool), developed during PhD project of Prof. An De Groef will be investigated. This clinical assessment tool consists of the assessment of soft-tissue adhesion at 7 locations at the upper limb region: axillary and breast region scars, pectoral region, axilla, frontal chest wall, lateral chest wall and the inframammary fold. At each location, the degree of the adhesions will be scored at three levels (skin, superficial and deep) on a 4-point scale (between no adhesions and very stiff adhesions).
  results will be compared with the results of the Myoton pro. approximately 1 week between test & retest
Validity of palpation for general stiffness | 1 week
  Palpation for general tissue stiffness scored on a Linkert Scale (0-5) at the different locations will be explored and the sum of total score of all locations will be calculated (0-35).
  results will be compared with the results of the Myoton pro. approximately 1 week between test & retest
Reliability for the assessment of movement functions | 1 week
  The reliability of goniometer, digital goniometer (EasyAngle®, Meloq AB, Stockholm) and inclinometer will be assessed for the following tasks: shoulder abduction, flexion, external rotation, and the ULIFT functional task. The inertial sensors are easy to use in daily practice, portable but come with a high cost in comparison to a goniometer, digital goniometer or inclinometer.
  The scapular movement assessment of the inertial sensors will be compared with the results of the inclinometer and digital goniometer. The glenohumeral movements will be compared with the results of the goniometer, digital goniometer and inclinometer.
  approximately 1 week between test & retest
Construct validity for the assessment of movement functions | 1 week
  The validity of goniometer, digital goniometer (EasyAngle®, Meloq AB, Stockholm) and inclinometer will be assessed for the following tasks: shoulder abduction, flexion, external rotation, and the ULIFT functional task. The inertial sensors are easy to use in daily practice, portable but come with a high cost in comparison to a goniometer, digital goniometer or inclinometer.
  The scapular movement assessment of the inertial sensors will be compared with the results of the inclinometer and digital goniometer. The glenohumeral movements will be compared with the results of the goniometer, digital goniometer and inclinometer.
  approximately 1 week between test & retest
Validity of machine learning model for Upper limb functioning from ActiGraph sensors for breast cancer survivors | 1 week
  The accelerometer to evaluate upper limb functioning will be validated against video annotated data as proposed by Lum and colleagues. Established methods use a machine learning pipeline to accurately and automatically recognize functional upper limb activities from accelerometer data in healthy subjects. These models will be evaluated against video annotated data to assess accuracy and correlation for our subsample of breast cancer survivors.
  approximately 1 week between test & retest
Validity of the use of hot/cold tubes for temperature sensations | 1 week
  Hot/cold tubes will be used for the cold and heat detection, but to validate this assessment method is will be compared with thermorollers.
  approximately 1 week between test & retest
Validity of the assessment of upper limb activities through accelerometry | 1 week
  The accelerometer will be used as comparable sign and dependent variable to evaluate the upper limb function to capture the 'activity and participation level' of the ICF model.
  approximately 1 week between test & retest
Validity of the assessment of upper limb activities: quickDASH | 1 week
  The quickDASH will be used as comparable sign and dependent variable to evaluate the upper limb function to capture the 'activity and participation level' of the ICF model.
  The QuickDASH is a shortened version of the DASH Outcome Measure. The QuickDASH uses 11 items to measure physical function and symptoms in people with any or multiple musculoskeletal disorders of the upper limb. The resultant score is reported on a scale of 0 to 100, where 0 represents no disability and 100 represents total disability
  approximately 1 week between test & retest

CONTACTS AND LOCATIONS:
Overall Officials: An De Groef, Prof. Dr., Principal Investigator — KU Leuven
Locations (1):
- Universitair Ziekenhuis Leuven, Leuven, Belgium

REFERENCES:
- [Background] De Groef A, Van der Gucht E, Dams L, Evenepoel M, Teppers L, Toppet-Hoegars J, De Baets L. The association between upper limb function and variables at the different domains of the international classification of functioning, disability and health in women after breast cancer surgery: a systematic review. Disabil Rehabil. 2022 Apr;44(8):1176-1189. doi: 10.1080/09638288.2020.1800835. Epub 2020 Aug 8. PMID 32772650
- [Background] De Groef A, Van Kampen M, Vervloesem N, De Geyter S, Dieltjens E, Christiaens MR, Neven P, Geraerts I, Devoogdt N. An evaluation tool for myofascial adhesions in patients after breast cancer (MAP-BC evaluation tool): Development and interrater reliability. PLoS One. 2017 Jun 9;12(6):e0179116. doi: 10.1371/journal.pone.0179116. eCollection 2017. PMID 28598978
- [Background] Yang EJ, Park WB, Seo KS, Kim SW, Heo CY, Lim JY. Longitudinal change of treatment-related upper limb dysfunction and its impact on late dysfunction in breast cancer survivors: a prospective cohort study. J Surg Oncol. 2010 Jan 1;101(1):84-91. doi: 10.1002/jso.21435. PMID 19924721
- [Background] Kilbreath SL, Refshauge KM, Beith JM, Ward LC, Lee M, Simpson JM, Hansen R. Upper limb progressive resistance training and stretching exercises following surgery for early breast cancer: a randomized controlled trial. Breast Cancer Res Treat. 2012 Jun;133(2):667-76. doi: 10.1007/s10549-012-1964-1. PMID 22286332
- [Background] Lum PS, Shu L, Bochniewicz EM, Tran T, Chang LC, Barth J, Dromerick AW. Improving Accelerometry-Based Measurement of Functional Use of the Upper Extremity After Stroke: Machine Learning Versus Counts Threshold Method. Neurorehabil Neural Repair. 2020 Dec;34(12):1078-1087. doi: 10.1177/1545968320962483. Epub 2020 Nov 5. PMID 33150830